CLINICAL TRIAL: NCT00037661
Title: Double-Masked, Randomized, Placebo-Controlled Study of Efficacy Parameter Following Administration of INS365 Ophthalmic Solution or Placebo in a Controlled Adverse Environment (CAE) Chamber in Subjects With Non-Sjogren's Associated Dry Eye
Brief Title: Study of INS365 Ophthalmic Solution in a Controlled Adverse Environment in Patients With Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-108
Record Dates: First submitted 2002-05-18; First posted 2002-05-20 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: dry eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

INTERVENTIONS:
Drug: INS365 Ophthalmic Solution

SUMMARY:
Comparative efficacy trial of INS365 Ophthalmic Solution and placebo in patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* have Non-Sjogren's associated dry eye disease with symptoms lasting greater than 6 months
* had intermittent or regular artificial tear use within past 3 months

Exclusion Criteria:

* had LASIK surgery
* had punctal occlusion or cauterization within last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2002-04; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)